CLINICAL TRIAL: NCT04631588
Title: Phase 1b Safety and Tolerability of Intradermal BOTOX® (OnabotulinumtoxinA) Purified Neurotoxin Complex in Participants With Facial Fine Lines
Brief Title: Intradermal (ID) BOTOX in the Treatment of Facial Fine Lines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1940-102-008
Record Dates: First submitted 2020-11-13; First posted 2020-11-17 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Facial Fine Lines
Keywords: Facial Fine Lines,BOTOX,Onabotulinum Toxin A
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Open Label BOTOX (Experimental): Participants will receive BOTOX at Baseline (Day 1)
  Interventions: Drug: Botox
- Double-Blind Randomized BOTOX (Experimental): Participants will receive BOTOX at Baseline (Day 1)
  Interventions: Drug: Botox
- Double Blind Randomized Placebo (Placebo Comparator): Participants will receive placebo at Baseline (Day 1)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botox — Intradermal (ID) injection
  Arms: Double-Blind Randomized BOTOX; Open Label BOTOX
Drug: Placebo — Intradermal (ID) injection
  Arms: Double Blind Randomized Placebo

SUMMARY:
The main objective of this study is to assess safety and tolerability of Intradermal (ID) BOTOX in participants with facial fine lines.

ELIGIBILITY:
Inclusion Criteria:

* A female participant must be willing to minimize the risk of inducing pregnancy for the duration of the clinical study (eg, for at least 90 days after receiving study intervention).
* Participant must have sufficient visual acuity without the use of eyeglasses (contact lans use acceptable) to accurately assess their facial lines, in the opinion of the investigator.
* Participant must be in good health as determined by medical history, physical examination, vital signs, and investigator's judgment, including no known active COVID-19 infection.
* Be nonsmoking and a nonuser of cannabis and nicotine-containing products, or have not smoked or used cannabis or nicotine-containing products, including e-cigarettes, within the previous 2 years.

Exclusion Criteria:

* Known immunization or hypersensitivity to any botulinum toxin serotype.
* Any medical condition that may put the participant at increased medical risk with exposure to BOTOX including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other condition that might interfere with neuromuscular function.
* Rosacea, skin infection, or any other skin disease or disorder that would represent a safety concern and/or interfere with the ability to either administer treatment or assess the treatment effect, as determined by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Baseline (Day 1) to Final Visit (up to Day 97)
  Unique number of participants who experience one or more treatment emergent adverse event
Number of Participants with Potential Clinically Significant (PCS) changes in vital signs | Baseline (Day 1) to Final Visit (up to Day 97)
  Unique number of participants who experience one or more Potential Clinically Significant (PCS) change in vital signs from the Baseline visit.
Number of Participants with Potential Clinically Significant (PCS) changes in physical exams | Baseline (Day 1) to Final Visit (up to Day 97)
  Unique number of participants who experience one or more Potential Clinically Significant (PCS) change in physical exams from the Baseline visit.
Number of Participants with injection site pain/discomfort. | Baseline (Day 1)
  Unique number of participants who experience injection site pain and/or discomfort at the injection site during administration of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (5):
- United States (5):
  - Skin and Cancer Associates, LLP /ID# 225152, Miami, Florida
  - Laser & Skin Surgery Center of New York /ID# 225153, New York, New York
  - Tennessee Clinical Research Center /ID# 225151, Nashville, Tennessee
  - Austin Institute for Clinical Research /ID# 225154, Pflugerville, Texas
  - Advanced Clinical Research /ID# 225155, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com.,To be considered as a site for current and future Allergan Clinical Trials, please register using the Investigator Databank link. — http://www.AllerganClinicalTrials.com